CLINICAL TRIAL: NCT07300943
Title: A Phase 1/2 Study of CLIO-8221 in Patients With Advanced Solid Tumors
Brief Title: Study in Advanced Solid Tumor Patients
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Callio Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CLIO-8221-001
Record Dates: First submitted 2025-12-14; First posted 2025-12-24 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Intervention Model Description: Phase 1: no randomization will be performed. Phase 2: participants in each cohort will be randomized with a 1:1 ratio to receive one of the expansion doses of CLIO-8221.
Masking Description: No, this is an open-label trial
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dose escalation and dose level expansion (Experimental): Phase 1: CLIO-8221 monotherapy in escalating doses. Phase 2: Phase 2 will be initiated in tumor-specific expansion cohorts at selected doses.
  Interventions: Drug: CLIO-8221

INTERVENTIONS:
Drug: CLIO-8221 — intravenous (IV) infusion

SUMMARY:
The study will be conducted in 2 phases: Phase 1: Dose-escalation and Dose Level Expansion, Phase 1 will determine the maximum tolerated dose (MTD) and/or recommended dose for expansion (RDE). Phase 2: Tumor-Specific Expansions with Dose Optimization, Phase 2 will further evaluate CLIO-8221 in tumor-specific expansion cohorts to optimize dosing and assess preliminary efficacy.

DETAILED DESCRIPTION:
Phase 1: Dose-escalation and Dose Level Expansion. Dose escalation safety data will be reviewed by a Safety Monitoring Committee (SMC) to guide dosing decisions. Backfill enrollment may be used to further characterize safety, PK/PD, and antitumor activity.

Phase 2: Tumor-Specific Expansions with Dose Optimization. Phase 2 will further evaluate CLIO-8221 in tumor-specific expansion cohorts to optimize dosing and assess preliminary efficacy. Safety, tolerability, PK/PD, and response data will support selection of the recommended Phase 2 dose (RP2D) for further development.

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced solid tumors
* Patients must have metastatic or unresectable disease not suitable for further local treatment and should have received prior beneficial therapies unless ineligible, unwilling, or lacking access.
* LVEF ≥50% by echocardiogram (ECHO) or multigated acquisition (MUGA) scan.
* An Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0 or 1
* Measurable disease per RECIST version 1.1 at baseline

Exclusion Criteria:

* Prior anti-tumor treatment with an ATRi.
* Prior or concurrent malignancy whose natural history or treatment has the potential to interfere with the safety or efficacy assessment of the investigational regimen. Exceptions are malignancies with a negligible risk of metastasis or death (e.g., 5-year OS ≥90%), including, but not limited to, adequately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, localized prostate cancer, ductal carcinoma in situ, and Stage I uterine cancer.
* History of uncontrolled seizure disorders or clinically significant neurodegenerative disorders, including progressive peripheral neuropathy. Stable Grade ≤ 2 peripheral neuropathy is allowed.
* Clinically significant autoimmune disease, either currently present or present within the previous 2 years, including a current requirement for systemic immunosuppressive therapy equivalent to >10 mg/prednisone daily (local immunosuppressive therapy such as inhaled or topical corticosteroids is allowed).
* Any uncontrolled Grade ≥ 3 (per NCI CTCAE version 6.0) viral, bacterial, or fungal infection within 2 weeks prior to Cycle 1 Day 1. Routine antimicrobial prophylaxis is permitted.
* History of hepatic cirrhosis, autoimmune hepatitis, or drug-associated hepatitis within the past 12 months.
* Uncontrolled diabetes mellitus, defined as Hgb A1c ≥8% or Hgb A1c between 7% and <8% with associated diabetes symptoms (polyuria or polydipsia) that are not otherwise explained.
* Any other medical, social, or psychosocial factors that, in the opinion of the investigator, could impact safety or compliance with study procedures.

Additional protocol defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Estimated)
Dates: Start 2026-02-28 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-07-17 (Estimated)

PRIMARY OUTCOMES:
Type, incidence, severity, and seriousness of adverse events (AEs) | Through end of treatment, up to approximately 2 years.
  Type, incidence, severity, and seriousness of AEs occurred
Type, incidence, and severity of laboratory abnormalities | Through end of treatment, up to approximately 2 years.
  Type, incidence, and severity of laboratory abnormalities occurred
Incidence of dose limiting toxicities dose (RP2D) of CLIO-8221 | From first dose through study day 21.
  Incidence of dose limiting toxicities occurred

SECONDARY OUTCOMES:
Objective Response Rate | Through disease progression, up to approximately 2 years.
  Participants who achieve partial or complete response per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria
Disease control rate | Through disease progression, up to approximately 2 years.
  Participants who achieve stable disease, partial or complete response per RECIST v1.1 criteria
Progression-free survival | Up to approximately 2 years.
  Time from first dose of CLIO-8221 to disease progression or death, whichever occurs first
Duration of objective response | From the date of enrollment until a confirmed partial or complete response is achieved, assessed up to 2 years.
  Time from the first documented objective tumor response (complete or partial), subsequently confirmed, to radiographic progression or death
Pharmacokinetic Parameter Area Under the Curve (AUC) for CLIO-8221 | Varying timepoints through end of treatment, up to approximately 2 years.
  Measure of CLIO-8221 AUC in plasma
Pharmacokinetic Parameter Maximum Concentration (Cmax) for CLIO-8221 | Varying timepoints through end of treatment, up to approximately 2 years.
  Measure of CLIO-8221 Cmax in plasma
Pharmacokinetic Parameter Time to Maximum Concentration (Tmax) for CLIO-8221 | Varying timepoints through end of treatment, up to approximately 2 years.
  Measure of CLIO-8221 Tmax in plasma
Pharmacokinetic Parameter Total Clearance (CL) for CLIO-8221 | Varying timepoints through end of treatment, up to approximately 2 years.
  Measure of CLIO-8221 CL in plasma
Pharmacokinetic Parameter Volume of distribution at steady state (Vd) for CLIO-8221 | Varying timepoints through end of treatment, up to approximately 2 years.
  Measure of CLIO-8221 Vd in plasma
Pharmacokinetic Parameter Apparent Terminal Half-life (t1/2) for CLIO-8221 | Varying timepoints through end of treatment, up to approximately 2 years.
  Measure of CLIO-8221 t1/2 in plasma

CONTACTS AND LOCATIONS:
Locations (10):
- United States (4):
  - DFCI, Boston, Massachusetts
  - MD Anderson Cancer Center, Houston, Texas
  - START San Antonio, San Antonio, Texas
  - START Mountain, West Valley City, Utah
- Australia (6):
  - Scientia Clinical Research, Randwick, New South Wales
  - Integrated Clinical Oncology Network Pty Ltd, South Brisbane, Queensland
  - Peter Maccallum Cancer Centre, Box Hill, Victoria
  - AlfredHealth, Heidelberg, Victoria
  - Royal Melbourne Hospital, Melbourne, Victoria
  - Linear Clinical Research Ltd, Nedlands, Western Australia

IPD SHARING:
Plan to Share IPD: No